CLINICAL TRIAL: NCT01060124
Title: Use of Durogesic D-TRANS in Cancer Pain Patients With Inadequately Controlled Pain Relief From Weak Opioids
Brief Title: An Efficacy and Safety Study of Transdermal Therapeutic System (TTS)-Fentanyl in Cancer Participants With Inadequately Controlled Pain by Non-Narcotic Analgesics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012256; FEN-KOR-13
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Pain; Cancer
Keywords: Pain; Cancer; TTS-Fentanyl D-trans; Durogesic D-trans
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal Therapeutic System (TTS)-Fentanyl D-trans (Experimental)
  Interventions: Drug: Fentanyl D-trans

INTERVENTIONS:
Drug: Fentanyl D-trans — Fentanyl D-trans will be applied as transdermal patch releasing drug at the rate of 12.5 microgram per hour (mcg/hr) for 3 days with a dose ranging from 12 mcg/hr to 50 mcg/hr.
  Other Names: Durogesic D-Trans

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Transdermal Therapeutic System (TTS)-fentanyl D-Trans (transdermal patch containing a drug that is put on the skin so the drug will enter the body through the skin) treatment in cancer participants of Korea with inadequately controlled pain by non-narcotic analgesics (drug used to control pain) and participant's satisfaction.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-arm, multicenter (conducted in more than one hospital or medical school team work on a medical research study), prospective (study following participants forward in time) study conducted to assess the efficacy and safety of TTS-fentanyl D-trans in cancer participants of Korea with inadequately controlled pain by non-narcotic analgesics and for participant's satisfaction. The participants will receive the initial dose of TTS-fentanyl D-trans patch releasing 12 micrograms per hour (12 mcg/hr) of fentanyl and will be increased by 12 mcg/hr or 25 mcg/hr, every 3 days depending on the participant's pain control. Efficacy will primarily be evaluated by participant's satisfaction with pain treatment. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who complains of cancer pain
* Participants who have taken non-opioid analgesics for the past one month for cancer pain relief purpose, but still have average 4 or higher pain level on the Visual Analogue Scale (VAS) for the last 24 hours
* Participants with an estimated life expectancy of at least 2 months
* Participants who are able to communicate with the investigator
* Participants who can avoid getting pregnant appropriately if there is a possibility of pregnancy during this study period

Exclusion Criteria:

* Participants participating in another clinical trial
* Participants with a history of oversensitive reaction to a narcotic analgesic or with an existing history of drug abuse
* Participants who have active skin disease, avoiding application of the transdermal system
* Participants with a history of CO2 (carbon di-oxide) retention (i.e. chronic obstructive pulmonary disease)
* Participants undergoing chemotherapy/radiotherapy right now or is going to get chemotherapy/radiotherapy within the study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Therapeutic System (TTS)-Fentanyl D-trans: Fentanyl D-trans was applied as transdermal patch releasing drug at the rate of 12.5 microgram per hour (mcg/hr) for 3 days with a dose ranging from 12 mcg/hr to 50 mcg/hr.
Period: Overall Study
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Started | 103
Completed | 66
Not Completed | 37
Not completed — Other | 16
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 103 participants, data for baseline characteristic (age) was available only for 98 participants.
  years | 60.81 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 103 participants, data for baseline characteristic (gender) was available only for 98 participants.
  Participants
    Female | 35
    Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Satisfied With Pain Treatment
Description: Participants were assessed for their satisfaction for pain treatment after the application of the Transdermal Therapeutic System (TTS)-fentanyl D-trans.
Time Frame: Day 29
Population: Per-Protocol (PP) analysis population included all participants who completed the clinical trial without violating the protocol among the participant who participated in the clinical trial.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Number analyzed (Participants) | 64
percentage of participants | 82.81 [73.57 to 92.06]

2. Secondary Outcome: Difference in Pain Intensity Before and After Administration of (TTS)-Fentanyl D-trans
Description: Pain intensity difference was measured by Visual Analog Scale (VAS) score, which ranges from 0 to 10 centimeter (cm) where 0 cm=no pain and 10 cm= unimaginably severe pain.
Time Frame: Day 1 and Day 29
Population: Full Analysis (FAS) population included all participants who meet the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Number analyzed (Participants) | 98
units on a scale
  Day 1 | 6.61 (1.62)
  Day 29 | 3.66 (2.42)

3. Other Pre Specified Outcome: Number of Participants With Detailed Reason for Satisfaction With the Pain Treatment
Description: Participants were assessed for satisfaction for pain treatment after the administration of the TTS-fentanyl D-trans in detail with satisfied reasons, which are excellent pain relieving effect, convenient administration, minor adverse event, generally satisfied and other.
Time Frame: Day 29
Population: Full Analysis (FAS) population included all participants who meet the inclusion and exclusion criteria. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Number analyzed (Participants) | 75
participants
  Excellent pain relieving effect | 32
  Convenient administration | 24
  Minor adverse event | 4
  Generally Satisfied | 15
  Other | 0

4. Other Pre Specified Outcome: Initial and End Point Dose of TTS-Fentanyl D-trans
Description: Dose of TTS-fentanyl D-trans were monitored at start and end of the trial.
Time Frame: Day 1 and Day 29
Population: Safety population included all participants who were administered the TTS-fentanyl D-trans at least once.
Measure: Mean (Standard Deviation); unit: microgram per hour (mcg/hr)
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Number analyzed (Participants) | 103
microgram per hour (mcg/hr)
  Initial dose | 12.00 (0.00)
  End-point dose | 26.47 (19.05)

5. Other Pre Specified Outcome: Number of Participants With Investigator's Overall Evaluation on the Pain Treatment
Description: Investigator assessed the participants for satisfaction on pain treatment after the administration of the TTS-fentanyl D-trans as very satisfied, satisfied, average, dissatisfied or very dissatisfied.
Time Frame: Day 29
Population: Full Analysis (FAS) population included all those participants who meet the inclusion and exclusion criteria. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Number analyzed (Participants) | 69
participants
  Very Satisfied | 16
  Satisfied | 43
  Average | 9
  Dissatisfied | 0
  Very Dissatisfied | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 29
Description: An adverse event may be an undesirable and unintended sign (including an abnormal measurement), symptom or disease which is related to the study drug in terms of time regardless of the existence of a causal relationship with the study drug.
Arm/Group | Transdermal Therapeutic System (TTS)-Fentanyl D-trans
Serious Adverse Events (participants affected / at risk) | 18/103
Other Adverse Events (participants affected / at risk) | 25/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS)-Fentanyl D-trans (N=103)
Death (General disorders) | 2
Pyrexia (General disorders) | 2
Disease Progression (General disorders) | 1
Abdominal distention (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Camptocormia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cerebral infraction (Cardiac disorders) | 1
Haemoglobin decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Cervical cord compression (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Therapeutic System (TTS)-Fentanyl D-trans (N=103)
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No